CLINICAL TRIAL: NCT01590420
Title: Cost-utility Study of CPAP Treatment in Obstructive Sleep Apnea Patients
Brief Title: Cost-utility Study of Continuous Positive Airway Pressure Treatment in Obstructive Sleep Apnea Syndrome Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Associação Fundo de Incentivo à Pesquisa (Other)
Responsible Party: Principal Investigator, Camila Furtado Rizzi, PhD, Associação Fundo de Incentivo à Pesquisa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Cost-utility of OSAS
Record Dates: First submitted 2012-05-01; First posted 2012-05-03 (Estimated); Last update posted 2012-05-03 (Estimated); Status verified 2012-05

CONDITIONS: Obstructive Sleep Apnea Syndrome
Keywords: OSA; Sleep; CPAP; Cost
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CPAP treatment (Experimental): 1000 patients with 3-years CPAP treatment after a PSG titration
  Interventions: Device: CPAP S8- Scape / Resmed

INTERVENTIONS:
Device: CPAP S8- Scape / Resmed — The pressure for treatment is according to PSG titration
  Other Names: S8 Escape; Resmed

SUMMARY:
The purpose of this study is to estimate the cost-utility of continuous positive airway pressure (CPAP) therapy in obstructive sleep apnea (OSA) patients in Sao Paulo city, Brazil, after 3 years of treatment and to estimate the cost-effectiveness of CPAP on the number of medical visits, hospitalizations, medical examinations, used medications, new case incidence and cost of traffic accidents and absence from work. It is also designed to estimate quality-adjusted extended years of life, and to assess cost-effects of the therapy (device, masks, supplies, maintenance/year for membership of professional consulting, electric power) on the cost-effectiveness

DETAILED DESCRIPTION:
OSA is highly prevalent in Sao Paulo city, Brazil. It is associated with significant comorbidities. The cost-utility study is important to (1) support decision-making on health policies, (2) to incorporate new technologies, (3) implementation of preventive programs and policy development assistance in the medical field.

Probably CPAP treatment in the long-term, will improve health, physical and mental state, and especially, reduces spending on public health, demonstrating cost-utility.

ELIGIBILITY:
Inclusion Criteria:

* Both genders
* Aged 30 to 70 years old
* AHI > 30 events/hour

Exclusion Criteria:

* Patients residing in other cities and states other than São Paulo / SP / Brazil
* Patients with no fixed residence
* Previous CPAP contact

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2011-03; Primary Completion 2011-03 (Actual); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
costs of medical events post CPAP treatment | 3 years
  To evaluate the health satuts costs post-CPAP treatment.
Number of hospitalizations | 3 years
Changes in medications | 3 years

SECONDARY OUTCOMES:
Costs relative to CPAP treatment | 3 years
  To evaluate the influence of CPAP device on directs health costs

CONTACTS AND LOCATIONS:
Overall Officials: Camila F Rizzi, PhD, Principal Investigator — Federal University of São Paulo; Dalva Poyares, PhD, Study Chair — Federal University of São Paulo; Sergio Tufik, PhD, Study Director — Federal University of São Paulo; Marcos F Bosi, PhD, Study Chair — Federal University of São Paulo
Locations (1):
- Associação Fundo de Incentivo à Pesquisa, São Paulo, São Paulo, Brazil